CLINICAL TRIAL: NCT07050576
Title: Deep Learning and Radiomics for Prediction of Lymph Node Metastasis in Early-stage Esophageal Squamous Cell Carcinoma
Brief Title: Lymph Node Metastasis in Early Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Early-ESCC-LNM-2024
Record Dates: First submitted 2025-06-26; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-09

CONDITIONS: ESCC; Lymph Node Metastasis; Radiomics
Keywords: ESCC; Lymph node metastasis; radiomics
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: A total of 400 patients with early-stage ESCC from our center were divided into training and test sets.
  Interventions: Diagnostic Test: The prediction model of lymph node metastasis in early esophageal squamous cell carcinoma
- B: A total of 100 patients with early-stage ESCC from other center were defined as external validation
  Interventions: Diagnostic Test: The prediction model of lymph node metastasis in early esophageal squamous cell carcinoma

INTERVENTIONS:
Diagnostic Test: The prediction model of lymph node metastasis in early esophageal squamous cell carcinoma — The predictive performance of the model was validated in the test set. The optimal prediction model was determined based on the AUC and ACC. To assess the robustness of the chosen model, ROC analysis was conducted on the external validation set.

SUMMARY:
This study aims to develop a predictive model using deep learning and radiomics to assess the likelihood of lymph node metastasis in patients with early-stage esophageal squamous cell carcinoma (ESCC). Lymph node metastasis is a critical factor in determining the treatment approach and prognosis for ESCC patients. By analyzing medical imaging data, we hope to create a non-invasive method that can assist doctors in making more accurate treatment decisions. This research could improve patient outcomes by enabling earlier and more tailored interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed early-stage (T1) ESCC
* Preoperative contrast-enhanced CT data within 2 weeks before surgery
* Without any treatment before surgical resection

Exclusion Criteria:

* Patients who underwent neoadjuvant therapy or endoscopic treatment
* Insufficient CT imaging or poor CT quality
* Incomplete pathology results
* Presence of metastatic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The radiomics features that affects the prediction of LNM in early-stage ESCC. All patients with early-stage ESCC from the hospitals
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
AUC(the area under the curve) values of the model | 4 years
  The performance and clinical relevance of the models were assessed by analyzing the area under the curve (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No